CLINICAL TRIAL: NCT04757740
Title: Autologous Platelet Rich Fibrin Versus Steroid in Ultrasound-Guided Sacroiliac Joint Injection for Joint Dysfunction (Randomized Comparative Study)
Brief Title: Comparison Between Platelet-rich Fibrin and Steroid for Intra-articular Injection for Sacroiliac Joint Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Amr hamdy Mahmoud, Assistant lecturer, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D240
Record Dates: First submitted 2021-02-14; First posted 2021-02-17 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain
Keywords: sacroiliac joint; platelet rich fibrin; ultrasound-guided
MeSH Terms: conditions — Low Back Pain | interventions — Lidocaine; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet rich fibrin Group (Active Comparator): Platelet rich fibrin. Group P
  Interventions: Biological: intra-articular Platelet rich fibrin and lidocaine
- Methylprednisolone acetate (Active Comparator): Group S
  Interventions: Drug: methylprednisolone acetate and lidocaine

INTERVENTIONS:
Biological: intra-articular Platelet rich fibrin and lidocaine — intra-articular injection of 3.5 ml of 1% lidocaine and PRF mixture.
  Other Names: Platelet rich fibrin Group
  Arms: Platelet rich fibrin Group
Drug: methylprednisolone acetate and lidocaine — intra-articular injection of Mixture of 40 mg of methylprednisolone acetate(1 ml) and 1% lidocaine (2.5 ml). intra-articular steroid
  Other Names: Steroid group
  Arms: Methylprednisolone acetate

SUMMARY:
Low back pain is one of the commonest complaints nowadays affecting nearly 20% of the population, Sacroiliac joint has been accused of being the primary cause of pain in about 10%: 27% of this population.

The sure diagnosis of sacroiliac joint pain is challenging because of multiple crossed factors of facet joint pain and intervertebral disc pain. Diagnosis can be done by history taking, local examination, imaging techniques, and controlled local anesthetic blocks.

Controlled local anesthetic blocks are diagnostic and therapeutic done by various methods either landmark-guided or imaging-assisted either by fluoroscopy, computed tomography (CT), magnetic resonance (MRI), or ultrasound-guided.

Lower cost, real-time viewing of needle leading to higher accuracy rate, and low ionizing radiation dose are favoring ultrasound-guided injection over other modalities.

Numerous treatment modalities are being used for sacroiliac joint pain ranging from physiotherapy and systemic analgesics like Non-steroidal anti-inflammatory drugs (NSAIDs) to minimally invasive intra-articular, periarticular injection, radiofrequency neurotomy, and surgical fusion of the joint.

Multiple injectates are being used for intraarticular injection most commonly local anesthetics and steroids which offer short-term symptomatic relief and delay the degenerative process.

The need for a longer duration effect directly affects the disease process itself aiming for accelerating the joint healing rate by biological growth factors found in human blood especially in platelets.

Platelet-rich plasma (PRP) has been used aiming to inject a high concentration of growth factors directly into the joint.

Platelet-rich fibrin (PRF), the second generation of platelet-rich plasma is now tried having the advantage of a simpler preparation and higher values of growth factors.

DETAILED DESCRIPTION:
Patient preparation:

History taking, physical examination, provocation tests (Gaenslen's test, Patrick's test, and Compression & distraction test), and investigations will be done according to the local protocol designed to evaluate these patients. This includes complete blood count, random blood glucose, serum creatinine & electrolytes, liver function tests, coagulation profile, and electrocardiogram (ECG).

Before the intervention, the participants will be informed about the visual analog scale (VAS) pain score (0-100 mm) (where 0=no pain and 100 = worst comprehensible pain) and the details of the procedures.

The patient will receive Midazolam 2 mg intravenous (IV) as a premedication. Intravenous access will be obtained with a 20-gauge intravenous (IV) cannula and monitors (pulse oximeter, electrocardiography, non-invasive blood pressure) will be applied.

We will use a high-frequency ultrasound probe .and a 22-gauge, 50 mm echogenic needle for performing the injection.

Injectable platelet-rich fibrin (iPRF) preparation:

blood collection will be done from the patient on the day of intervention in a 9 ml blank tube. Within maximum 2:3minutes from sampling, it will be placed in the horizontal centrifuge for a low-speed centrifuge for 8 minutes at 600 rpm 44 g. Upon termination of this process, the Orange color area in the tube (i-PRF) and the remaining blood materials below will be noticed. Then, the tubes will be opened cautiously to avoid remixing, 2.5 ml of i-PRF will be collected from the tubes using a 5ml syringe.

Ultrasound-guided technique:

The patient will be positioned in a prone position over a cushion and after -sterilization with povidone-iodine and draping, the probe will be positioned transversely over the 5th lumber spinous process then moving the probe downwards until sacrum can be identified. Then moving the probe slightly lateral till identifying the 1st posterior sacral foramina (seen as a break in the hyperechoic contour of the sacral wing) then moving the probe downwards till the 2nd posterior sacral foramina will be identified. Tilting the lateral part of the probe slightly upwards and visualizing lateral sacral crest, sacroiliac joint, and iliac bone. Using color Doppler to ensure the absence of vascularization at the injection site of the joint (if present moving the probe cranially or caudally until disappearance). after anesthetizing the skin with 2 ml of 2% lidocaine, the needle will be advanced in-plane to the joint and 0.1 ml of sterile water will be injected to ensure spread into sacroiliac joint by unidirectional flow with Color Doppler box then the 3.5 ml of 1% lidocaine and PRF mixture will be injected in the group (P) or 40 mg of methylprednisolone acetate (Depo-Medrol, Pfizer) (1 ml) and 1% lidocaine (2.5 ml) in the group (S).

Post-procedural care:

The Patient will be transferred to post-intervention care unit for 2 hours after the procedure monitoring heart rate, oxygen saturation, and any possible adverse effect then patients will be discharged to home with a prescription of Diclofenac potassium 50 mg tab three times daily (TID), diclofenac diethylamine gel topically TID and baclofen 10 mg tab TID.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged >18 years with Low back pain > 6 months.
2. Failure of conservative treatment for 3 months.
3. Positive findings on at least one of three provocation tests for sacroiliac joint pain: Gaenslen's test, Patrick's test, and compression & distraction test.
4. Positive diagnostic injection (pain reduction >80% after injection).

Exclusion Criteria:

1. Patient refusal.
2. Disorders in the hip joint.
3. Signs of lumbar radiculopathy.
4. Bleeding disorders including anticoagulation medications.
5. Positive response to Kemp's test (pain provocation test for sciatica).
6. Infection at site of injection.
7. Psychiatric problems as prevent completion of the study related questionnaires.
8. Morbid obesity BMI > 40.
9. Severe cardiac and respiratory disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment by VAS score | 1 month after procedure
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain

SECONDARY OUTCOMES:
Pain assessment by VAS score | 5 minutes after procedure
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
Pain assessment by VAS score | 1 week after procedure
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
Pain assessment by VAS score | 3 month after procedure
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
Pain assessment by VAS score | 6 month after procedure
  the quality of analgesia between (0-100 mm) where 0=no pain and 100 = worst comprehensible pain
Modified Oswestry Disability Index | 1 month after procedure
  to assess level of disability.
Modified Oswestry Disability Index | 6 month after procedure
  to assess level of disability.
Patient satisfaction with procedure | 1 month after procedure
  Will be evaluated according to a satisfaction score (poor = 0; fair = 1; good = 2; excellent= 3)
patient discomfort with procedure | 5 minutes after procedure
  yes or no question
hematoma | 5 minutes after procedure
  procedure related complication
Allergy | 10 minutes after procedure
  procedure related complication
Age | 5 minutes before procedure
  In years
weight | 5 minutes before procedure
  In kilograms
Height | 5 minutes before procedure
  In meters
BMI | 5 minutes before procedure
  In kilogram per square meter
Analgesic requirement after injection | 1 day after procedure
  analgesic dose needed after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Alsaeid, MD, Study Director — Fayoum University Hospitals
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt